CLINICAL TRIAL: NCT04691583
Title: Study on the Mechanism of Regulating Gut Microbiome in Obese People by Regulating Brain-gut Axis With Fast Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20180520
Record Dates: First submitted 2020-12-27; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Obesity; Gastrointestinal Microbiome; Magnetic Resonance Imaging
Keywords: Obesity；Gut microbiome；Task fMRI;Brain-Gut axis
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: 1. Normal diet：Starting from May 20, 2018, the subjects will eat a normal diet for 4 days, with no restriction on calories and food types. The subjects are required to record their daily diet and dietary intake of calories.
  2. Fast diet of High control ：From May 24, 2018, the method of fast diet was adopted on alternate days. According to the dietary records of normal diet, the normal caloric intake of each subject was calculated. Fast diet was carried out according to 2/3, 1/2, 1/3 and 1/4 of the original normal caloric intake.Each caloric stage last for 4 days, and the total cycle of fast diet was 31 days.
  3. Fast diet of Low control ：After the intervention of fast diet of high control, the subjects were allowed to continue the diet fast diet every other day. It was suggested that the daily caloric intake was 600kal/ day for males and 500kal/ day for females.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fast diet — Fast diet of High control ：From May 24, 2018, the method of fast diet was adopted on alternate days. According to the dietary records of normal diet, the normal caloric intake of each subject was calculated. Fast diet was carried out according to 2/3, 1/2, 1/3 and 1/4 of the original normal caloric intake.Each caloric stage last for 4 days, and the total cycle of fast diet was 31 days.
  Fast diet of Low control ：After the intervention of fast diet of high control, the subjects were allowed to continue the diet fast diet every other day. It was suggested that the daily caloric intake was 600kal/ day for males and 500kal/ day for females.

SUMMARY:
1. Normal diet：Starting from May 20, 2018, the subjects will eat a normal diet for 4 days, with no restriction on calories and food types. The subjects are required to record their daily diet and dietary intake of calories.
2. Fast diet of High control ：From May 24, 2018, the method of fast diet was adopted on alternate days. According to the dietary records of normal diet, the normal caloric intake of each subject was calculated. Fast diet was carried out according to 2/3, 1/2, 1/3 and 1/4 of the original normal caloric intake.Each caloric stage last for 4 days, and the total cycle of fast diet was 31 days.
3. Fast diet of Low control ：After the intervention of fast diet of high control, the subjects were allowed to continue the diet fast diet every other day. It was suggested that the daily caloric intake was 600kal/ day for males and 500kal/ day for females.

DETAILED DESCRIPTION:
1. Normal diet: the course of treatment was 4 days. The subjects were asked to record the daily diet and dietary intake in the daily observation scale (Table 1).
2. High control diet intervention: the course of treatment was 31 days. According to the actual intake of calories, 2 / 3, 1 / 2, 1 / 3 and 1 / 4 of the actual intake of the subjects were calculated as the light fasting calories. The treatment course of each calorie stage was 4 days. The subjects recorded the daily diet and dietary intake, and the nutritionists calculated the daily calorie intake and dietary types of each subject according to the daily calorie intake of each subject's normal diet. During the period of high control diet intervention, the diet on the day of light fasting was provided by the research group. Besides the diet provided by the research group, other foods (except water without calories) were strictly prohibited on the day of light fasting.
3. Low control diet intervention: the course of treatment was 31 days. It is suggested that the calorie intake of men and women should be 600 kcal / day and 500 kcal / day on the day of light fasting. The diet type can refer to the recipe made by the nutritionist.

ELIGIBILITY:
Inclusion Criteria:

1. BMI greater than or equal to 28 kg/m2, waist circumference greater than or equal to 90cm for men and 85cm for women.
2. Aged between 18 and 60.
3. Patients may be accompanied by diseases such as abnormal blood pressure, abnormal blood lipid, abnormal uric acid, metabolic syndrome, respiratory sleep, constipation, etc., but they can only participate in these diseases if there is no obvious risk after clinical evaluation.
4. No serious heart, brain, liver and kidney dysfunction, uremia coma, ketoacidosis, hypoglycemia, anemia, malnutrition, hematopoietic system and body immune system diseases, infectious diseases, neurological diseases.

5, the body does not contain the implantation or other metal materials such as the implantable metal denture, cardiac pacemaker, artificial joint, insulin pump and so on, no claustrophobia, non-pregnancy, suitable for magnetic resonance examination to participate in.

Exclusion Criteria:

1. those who do not meet the above diagnostic criteria have poor compliance and have not signed a voluntary informed consent to participate in the experimental study.
2. patients with severe cardiac, cerebral, hepatic and renal dysfunction, uremia coma, ketoacidosis, hypoglycemia, anemia, malnutrition, hematopoietic system and physical immune system diseases, infectious diseases, neurological diseases, etc.
3. special groups such as female menstruation, minors, pregnant women, and the elderly over 60 years old.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
ReHo | 1 month
  Reho of brain after 1 month of fast diet
ReHo | 2 month
  Reho of brain after 2 month of fast diet
Adiponectin | 1 month
  Adiponectin after 1 month of fast diet
Adiponectin | 2 month
  Adiponectin after 2 month of fast diet
Gut microbiome | 1 month
  the change of gut microbiome after 1 month of fast diet
Gut microbiome | 2 month
  the change of gut microbiome after 2 month of fast diet
body mass | 1 month
  the change of body mass after 1 month of fast diet
body mass | 2 month
  the change of body mass after 2 month of fast diet

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No